CLINICAL TRIAL: NCT06331442
Title: The Effect of Photodynamic Therapy on Accumulation and Bacteriological Composition of Dental Plaque in Orthodontic Patients
Brief Title: The Effect of Photodynamic Therapy on Plaque in Orthodontic Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Tadeja Blagec, Doctor of Dental Medicine, University of Zagreb
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 006503905
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Plaque, Dental; Dental Plaque Induced Gingivitis; White Spot Lesion
Keywords: dental plaque; gingiva; white spot lesion; photodynamic therapy; chlorhexidine varnish; tricalcium phosphate varnish; fluoride
MeSH Terms: conditions — Dental Plaque | interventions — Photochemotherapy; tricalcium phosphate; tenocyclidine; Paint

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Photodynamic therapy group (Experimental): Group of participants (n=10) allocated to this group will receive photodynamic therapy which consists of toluidine blue based dye (155 mg/mL) and 660 nm diode laser. Participants will be subjected to this treatment right after the placement of a fixed orthodontic appliance (T0), 6 weeks (T1) and 12 weeks (T2) later.
  Interventions: Other: Photodynamic therapy
- Tricalcium phosphate varnish with 5% NaF group (Active Comparator): Group of participants (n=10) allocated to this group will receive tricalcium varnish with 5% NaF which will be applied according to the manufacturer's recommendations. Participants will be subjected to this treatment right after the placement of a fixed orthodontic appliance (T0), 6 weeks (T1) and 12 weeks (T2) later.
  Interventions: Other: Tricalcium phosphate (TCP) varnish with 5% NaF
- Chlorhexidine varnish group (Active Comparator): Group of participants (n=10) allocated to this group will receive chlorhexidine varnish which will be applied according to the manufacturer's recommendations. Participants will be subjected to this treatment right after the placement of a fixed orthodontic appliance (T0), 6 weeks (T1) and 12 weeks (T2) later.
  Interventions: Other: Chlorhexidine varnish
- Negative control group (No Intervention): Group of participants (n=10) allocated to this group will not receive an intervention.

INTERVENTIONS:
Other: Photodynamic therapy — Patients allocated to the first group (n=10) will receive photodynamic therapy. Buccal/labial surface around the bracket of each tooth in the upper dental arch (from right to left second premolar) will be treated with toluidine blue based dye (155 mg/mL; LaserHF Paro-PDT, Hager & Werken, GmbH & Co. Kg, Duisburg, Germany). This photosensitive solution will be applied on teeth with the sterile syringe and left for 60 s. Then, the excess of the photosensitive solution will be rinsed with the sterile syringe containing a saline solution. Then, a 660 nm diode laser (Laser HF, Hager & Werken, GmbH & Co. Kg, Duisburg, Germany) will be used for photoactivation (power output 100 mW, power density 124.34 W/cm2 and continuous working mode). Buccal/labial surface of each tooth will be radiated for 60 s at approximately 5 mm away from the enamel surface. This intervention will be performed right after the placement of a fixed orthodontic appliance (T0), 6 weeks (T1) and 12 weeks (T2) later.
  Arms: Photodynamic therapy group
Other: Tricalcium phosphate (TCP) varnish with 5% NaF — Tricalcium phosphate varnish with 5% NaF (Clinpro™ White Varnish, 3M ESPE 3M Deutschland GmbH, Germany) will be applied to the patients allocated to the second group (n=10). The varnish will be applied to the buccal/labial surfaces of 10 teeth in the upper dental arch (from right to left second premolar) according to the manufacturer's recommendations. This intervention will be performed right after the placement of a fixed orthodontic appliance (T0), 6 weeks (T1) and 12 weeks (T2) later.
  Arms: Tricalcium phosphate varnish with 5% NaF group
Other: Chlorhexidine varnish — Chlorhexidine varnish (1% CHX, 1% thymol; Cervitec® Plus, Ivoclar Vivadent AG, Schaan, Liechtenstein) will be applied to the patients allocated to the third group (n=10). The varnish will be applied to the buccal/labial surfaces of 10 teeth in the upper dental arch (from right to left second premolar) according to the manufacturer's recommendations. This intervention will be performed right after the placement of a fixed orthodontic appliance (T0), 6 weeks (T1) and 12 weeks (T2) later.
  Arms: Chlorhexidine varnish group

SUMMARY:
This randomized controlled trial will be conducted on 40 orthodontic patients at the Department of Orthodontics, University Hospital Centre Zagreb, Croatia. Respondents will be randomly allocated into 4 groups (n=10). The first group will receive photodynamic therapy, the second tricalcium phosphate varnish with 5% NaF (sodium fluoride), the third 1% chlorhexidine varnish, while the fourth group will be the negative control. Before and after the mentioned interventions, the participants will have the amount of plaque measured using the plaque index and the bacteriological composition of the plaque assessed using the mass spectrometry and PCR. The gingival condition will be assessed using the gingival index. Also, the occurrence of white spot lesions will be evaluated on intraoral photographs.

DETAILED DESCRIPTION:
Goals of this research are: 1. To compare the plaque index in orthodontic patients treated with different antibacterial agents (photodynamic therapy, tricalcium phosphate varnish with 5% NaF, chlorhexidine varnish) before insertion of a fixed orthodontic appliance (T0), 6 weeks (T1), 12 weeks (T2) and 18 weeks later (T3); 2. To compare the bacteriological composition of supragingival plaque using the mass spectrometry in orthodontic patients treated with different antibacterial agents before insertion of a fixed orthodontic appliance (T0), 6 weeks (T1), 12 weeks (T2) and 18 weeks later (T3); 3. To compare the bacteriological composition of subgingival plaque using polymerase chain reaction in orthodontic patients treated with different antibacterial agents before insertion of a fixed orthodontic appliance (T0) and 18 weeks later (T3); 4. To compare the gingival index in orthodontic patients treated with different antibacterial agents before insertion of a fixed orthodontic appliance (T0), 6 weeks (T1), 12 weeks (T2) and 18 weeks later (T3); 5. To compare the occurrence of white spot lesions in orthodontic patients treated with different antibacterial agents before insertion of a fixed orthodontic appliance (T0) and 18 weeks later (T3).

This study hypothesizes that photodynamic therapy is just as effective in reducing plaque accumulation, reducing bacteria in supragingival and subgingival plaque, preventing gingival inflammation and preventing initial carious lesions (white spot lesions) in orthodontic patients as tricalcium phosphate varnish with 5% NaF and 1% chlorhexidine varnish.

Participants (40 orthodontic patients at the Department of Orthodontics, University Hospital Centre Zagreb, Croatia) will be randomly assigned to one of four groups. Randomization will be performed before the recruitment using software for randomization (Research Randomizer; permuted blocks randomization). Outcome assessor will be blinded, while participants and care providers will be aware of the group allocation.

Group of participants (n=10) allocated to the first group will receive photodynamic therapy which consists of toluidine blue based dye (155 mg/mL) and 660 nm diode laser. Participants (n=10) allocated to the second group will receive tricalcium varnish with 5% NaF which will be applied according to the manufacturer's recommendations. Group of participants (n=10) allocated to the third group will receive chlorhexidine varnish which will be applied according to the manufacturer's recommendations. All interventions will be performed right after the placement of a fixed orthodontic appliance (T0), 6 weeks (T1) and 12 weeks (T2) later. The fourth group (n=10) will be the negative control which means that participants will not receive any intervention.

Primary outcome measures: assessment of dental plaque accumulation using plaque index and assessment of the bacteriological composition of supragingival plaque using mass spectrometry. Secondary outcome measures: assessment of the bacteriological composition of subgingival plaque using the polymerase chain reaction, assessment of gingival condition using the gingival index and diagnosis of white spot lesions on intraoral photographs.

ELIGIBILITY:
Inclusion Criteria:

* 12 to 17 years of age
* indication for fixed orthodontic treatment without the need for extraction
* permanent dentition (including second molars)
* absence of oral lesions, caries, pulpal and periapical diseases and gingival and periodontal diseases

Exclusion Criteria:

* previous orthodontic treatment
* taking antibiotics and anti-inflammatory drugs 3 months before the study and during the study
* use of antiseptic rinses 3 months before the study and during the study
* taking corticosteroids and immunosuppressive drugs
* smoking
* systemic conditions that can affect the inflammatory response of soft tissues and the possibility of maintaining adequate plaque control (diabetes, immune disorders, etc.)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Assessment of dental plaque accumulation using plaque index | 18 weeks
  In T0, plaque accumulation on upper 10 teeth (from right to left second premolar) will be measured using Silness and Löe plaque index.
  In T1, T2 and T3 the accumulation of plaque will be measured using the modified Silness and Löe plaque index. The plaque index will be measured on the upper 10 teeth (from right to left second premolar). The tooth surface around the bracket will be divided into 4 areas - mesial, distal, gingival and occlusal. In each area, the level of plaque will be expressed on a scale from 0 to 3: 0- no dentobacterial plaque; 1- flecks of dentobacterial plaque; 2- continuous line of dentobacterial plaque≤1 mm; 3- continuous line of dentobacterial plaque>1 mm. Plaque index will be measured before insertion of a fixed orthodontic appliance (T0), 6 weeks (T1), 12 weeks (T2) and 18 weeks later (T3).
Assessment of the bacteriological composition of supragingival plaque using mass spectrometry | 18 weeks
  A sample of supragingival plaque will be taken from all 10 examined teeth in the upper dental arch using a sterile probe. The sample will be stored in an Eppendorf plastic tube containing 1.5 mL of physiological solution. From the solution, 0.01 μL of the sample will be inoculated onto blood/Brucella and Columbia agar and incubated aerobically and anaerobically. After incubation, visible bacterial colonies will be counted in CFU (colony forming units) and identified by the MALDI-TOF (matrix assisted laser desorption/ionization) method. A sample for microbiological analysis will be taken before insertion of a fixed orthodontic appliance (T0), 6 weeks (T1), 12 weeks (T2) and 18 weeks later (T3).

SECONDARY OUTCOMES:
Assessment of the bacteriological composition of subgingival plaque using polymerase chain reaction | 18 weeks
  A sample of subgingival plaque will be taken from the gingival sulcus of all 10 examined teeth in the upper dental arch using sterile paper points (#50). The paper point will be placed in the gingival sulcus up to 4 mm or until resistance is felt and left for 20-30 seconds. After that, the paper point with the sample will be placed in an Eppendorf plastic tube containing 1.5 mL of physiological solution and will be stored at -80 ℃. The samples will then be analyzed by the molecular method- polymerase chain reaction. Primers will be used to detect the following bacteria: Aggregatibacter actynomicetemcomitans, Porphyromonas gingivalis, Porphyromonas endodontalis, Treponema denticola, Tannerella forsythia and Fusobacterium nucleatum. A sample for molecular analysis will be taken before insertion of a fixed orthodontic appliance (T0) and 18 weeks later (T3).
Assessment of gingival condition using gingival index | 18 weeks
  The gingival condition will be assessed using Silness and Löe gingival index on 10 teeth in the upper dental arch (from right to left second premolar). The soft tissue around the tooth will be divided into 4 parts/areas: distolabial/buccal papilla, labial marginal gingiva, mesiolabial/buccal papilla, and palatal marginal gingiva. In each area, inflammation of the gingiva will be expressed on a scale from 0 to 3, as follows: 0- normal gingiva; 1- mild inflammation- slight change in color, slight oedema, no bleeding on probing; 2- moderate inflammation- redness, oedema and glazing, bleeding on probing; 3- severe inflammation- marked redness and oedema, ulceration, tendency to spontaneous bleeding. Gingival index will be measured before insertion of a fixed orthodontic appliance (T0), 6 weeks (T1), 12 weeks (T2) and 18 weeks later (T3).
Diagnosis of white spot lesions on intraoral photographs | 18 weeks
  The labial surfaces of 10 teeth in the upper dental arch (from right to left second premolar) will be photographed. Intraoral photographs (frontal, left and right sagittal) will be taken using a camera (Nikon digital camera d7500, Nikon, Tokio, Japan) at settings ISO=125, f=32. The photos taken in the first and last visit will be placed next to each other on the monitor and compared. An identical white spot lesion on photographs taken at T0 and T3 (same size and surface) will be considered a developmental or fluoride white spot. A white spot that was present at T0 but worsened (enlarged spot or changed surface) over time will be recorded as a white spot lesion. Photographs will be taken before insertion of a fixed orthodontic appliance (T0) and 18 weeks later (T3).

CONTACTS AND LOCATIONS:
Overall Officials: Tadeja Blagec, DMD, Principal Investigator — University of Zagreb

REFERENCES:
- [Derived] Blagec T, Simunovic L, Budimir A, Gabric D, Mestrovic S. The influence of photodynamic therapy on the supragingival plaque accumulation and bacterial composition in orthodontic patients: a randomized controlled trial. Eur J Orthod. 2025 Sep 17;47(5):cjaf072. doi: 10.1093/ejo/cjaf072. PMID 41091662